CLINICAL TRIAL: NCT01330589
Title: The Effect of Inducing the Cytochrome P450 System on the Pharmacodynamic Efficacy of Clopidogrel
Brief Title: Pharmacodynamic Study on Efficacy of Clopidogrel With St. John's Wort
Acronym: INDUCE-it
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll subjects and changes in standard of care for PCI
Sponsor: Lancaster General Hospital (Other)
Collaborators: H G Barsumian MD Memorial Fund (Other); Louise von Hess Medical Research Institute (Other)
Responsible Party: Principal Investigator, Michael A. Horst, PhD, MPHS, MS, Director of Research, Lancaster General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-56-LGH
Record Dates: First submitted 2011-03-28; First posted 2011-04-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Percutaneous coronary intervention; Clopidogrel; St. John's Wort; CYP 2C19 loss-of-function allele
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AB: Placebo (A); St. Johns Wort (B) (Experimental): Receive placebo for 7 days, 7 days washout and 7 days of St. Johns Wort
  Interventions: Drug: Placebo; Drug: St. Johns Wort
- BA: St. Johns Wort (B); Placebo (A) (Experimental): Receive St. Johns Wort for 7 days, 7 days washout and 7 days of placebo
  Interventions: Drug: Placebo; Drug: St. Johns Wort

INTERVENTIONS:
Drug: Placebo — Non-active placebo for 7 days: PO/TID
Drug: St. Johns Wort — For 7 days: 300mg PO/TID

SUMMARY:
The purpose of this study is to evaluate whether patients post PCI receiving clopidogrel who are carriers of at least one CYP 2C19 loss-of-function allele may achieve improved pharmacodynamic efficacy of clopidogrel when treated with the CYP 2C19 enzyme inducing agent, St. John's wort, as compared with placebo.

Hypothesis

1. Reduced platelet reactivity is present in patients receiving St. John's wort as compared to placebo when utilized in combination with clopidogrel
2. The combination or St. John's wort and clopidogrel results in enhanced platelet inhibition

DETAILED DESCRIPTION:
Objective The purpose of this study is to evaluate whether patients post PCI receiving clopidogrel who are carriers of at least one CYP 2C19 loss-of-function allele may achieve improved pharmacodynamic efficacy of clopidogrel when treated with the CYP 2C19 enzyme inducing agent, St. John's wort, as compared with placebo.

Specific Aims

1. To identify the difference in platelet reactivity in patients receiving St. John's wort or placebo
2. To characterize the difference in platelet inhibition in patients receiving St. John's wort or placebo

Hypothesis

1. Reduced platelet reactivity is present in patients receiving St. John's wort as compared to placebo when utilized in combination with clopidogrel
2. The combination or St. John's wort and clopidogrel results in enhanced platelet inhibition

Study Design The study is a prospective, randomized, double-blind, placebo-controlled, cross-over study of patients post PCI who require dual-antiplatelet therapy with aspirin and clopidogrel. Approximately 84 patients will be enrolled and undergo pharmacogenetic testing to assess clopidogrel responsiveness utilizing CYP P450 2C19 genotyping (Plavitest®). Based upon an assumption of 30% genetic non-responsiveness and a dropout rate of 20%, to achieve a final sample size of 20 subjects in the randomized crossover portion of the study, the investigators need to enroll approximately 84 subjects. Patients identified as carriers of at least one CYP 2C19 loss-of-function allele (i.e. clopidogrel reduced-metabolizers) will remain in the study and be randomly assigned to receive placebo or St. John's wort. Patients not carrying a CYP 2C19 loss-of-function allele (i.e. clopidogrel normal metabolizers) will not require any further follow-up as these patients are considered to display a normal response to clopidogrel. On day 7 following the initiation of the study drug, platelet function testing will be performed. Following a 7 day washout period, patients will be crossed over into the other study group to receive 7 days of study medication. On day 21, the patients will undergo platelet function testing and the study medication will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older
* Patients with a history of ACS and/or who receive PCI with stent placement at Lancaster General Hospital requiring dual antiplatelet therapy with aspirin and clopidogrel.

Exclusion Criteria:

* Patients with active or any known history of bleeding such as gastrointestinal, intracranial, or any other bleeding diathesis
* History of major surgery in the last year (any surgical procedure that involves general anesthesia or respiratory assistance)
* Clinical findings associated with an increased risk of bleeding at the judgment of the investigator
* Patients actively receiving anticoagulation therapy
* Hemoglobin < 10 g/dL
* Platelets < 150,000/mm3
* Known hepatic dysfunction
* History of intracranial malignancy or stroke
* Patients receiving thienopyridines chronically prior to PCI
* Concurrent use of CYP P450 2C19 substrates, or inhibiting/ inducing medications with the exception of proton pump inhibitors
* Illicit drug or alcohol abuse
* Daily treatment with nonsteroidal anti-inflammatory drugs or cyclooxygenase-2 inhibitors
* Allergy to St. Johns wort or lactose
* Patients expected to discontinue dual antiplatelet therapy prior to completion of the study protocol
* Patients unable to adhere to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean platelet reactivity (as measured in platelet reactivity units) on day 7 and day 21 | Day 7 and Day 21
  The investigators are comparing the mean platelet reactivity (as measured in platelet reactivity units) within subjects (treatment effect) between placebo and St. Johns Wort. In addition we will be assessing the period effect (difference between those getting treatment AB - placebo/St. Johns Wort and those getting treatment BA - St. Johns Wort/placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Kathy M Makkar, PharmD, Principal Investigator — Lancaster General Hospital; Roy S Small, MD, Principal Investigator — Lancaster General Hospital; Rupal P Dumasia, MD, Principal Investigator — Lancaster General Hospital; Jill A Rebuck, PharmD, Principal Investigator — Lancaster General Hospital; Michael A Horst, PhD, Principal Investigator — Lancaster General Research Institute; Yee M Lee, PharmD, Principal Investigator — Lancaster General Hospital; Richard D Paoletti, RPh, Principal Investigator — Lancaster General Hospital
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

REFERENCES:
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Steinhubl SR, Berger PB, Mann JT 3rd, Fry ET, DeLago A, Wilmer C, Topol EJ; CREDO Investigators. Clopidogrel for the Reduction of Events During Observation. Early and sustained dual oral antiplatelet therapy following percutaneous coronary intervention: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2411-20. doi: 10.1001/jama.288.19.2411. PMID 12435254
- [Background] Bhatt DL, Fox KA, Hacke W, Berger PB, Black HR, Boden WE, Cacoub P, Cohen EA, Creager MA, Easton JD, Flather MD, Haffner SM, Hamm CW, Hankey GJ, Johnston SC, Mak KH, Mas JL, Montalescot G, Pearson TA, Steg PG, Steinhubl SR, Weber MA, Brennan DM, Fabry-Ribaudo L, Booth J, Topol EJ; CHARISMA Investigators. Clopidogrel and aspirin versus aspirin alone for the prevention of atherothrombotic events. N Engl J Med. 2006 Apr 20;354(16):1706-17. doi: 10.1056/NEJMoa060989. Epub 2006 Mar 12. PMID 16531616
- [Background] Kimura T, Morimoto T, Kozuma K, Honda Y, Kume T, Aizawa T, Mitsudo K, Miyazaki S, Yamaguchi T, Hiyoshi E, Nishimura E, Isshiki T; RESTART Investigators. Comparisons of baseline demographics, clinical presentation, and long-term outcome among patients with early, late, and very late stent thrombosis of sirolimus-eluting stents: Observations from the Registry of Stent Thrombosis for Review and Reevaluation (RESTART). Circulation. 2010 Jul 6;122(1):52-61. doi: 10.1161/CIRCULATIONAHA.109.903955. Epub 2010 Jun 21. PMID 20566955
- [Background] Savi P, Herbert JM, Pflieger AM, Dol F, Delebassee D, Combalbert J, Defreyn G, Maffrand JP. Importance of hepatic metabolism in the antiaggregating activity of the thienopyridine clopidogrel. Biochem Pharmacol. 1992 Aug 4;44(3):527-32. doi: 10.1016/0006-2952(92)90445-o. PMID 1510701
- [Background] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Wang LS, Zhu B, Abd El-Aty AM, Zhou G, Li Z, Wu J, Chen GL, Liu J, Tang ZR, An W, Li Q, Wang D, Zhou HH. The influence of St John's Wort on CYP2C19 activity with respect to genotype. J Clin Pharmacol. 2004 Jun;44(6):577-81. doi: 10.1177/0091270004265642. PMID 15145964
- [Background] Barnes PM, Powell-Griner E, McFann K, Nahin RL. Complementary and alternative medicine use among adults: United States, 2002. Adv Data. 2004 May 27;(343):1-19. PMID 15188733
- [Background] Wang LS, Zhou G, Zhu B, Wu J, Wang JG, Abd El-Aty AM, Li T, Liu J, Yang TL, Wang D, Zhong XY, Zhou HH. St John's wort induces both cytochrome P450 3A4-catalyzed sulfoxidation and 2C19-dependent hydroxylation of omeprazole. Clin Pharmacol Ther. 2004 Mar;75(3):191-7. doi: 10.1016/j.clpt.2003.09.014. PMID 15001970
- [Background] Lau W, Carville D, Guyer K, Neer C. St. John's wort enhances the platelet inhibitor effect of clopidogrel in clopidogrel "resistant" healthy volunteers. J Am Coll Cardiol 2005;4:382A(abstract).
- [Background] Lau WC, Welch TD, Shields T, Rubenfire M, Tantry US, Gurbel PA. The effect of St John's Wort on the pharmacodynamic response of clopidogrel in hyporesponsive volunteers and patients: increased platelet inhibition by enhancement of CYP3A4 metabolic activity. J Cardiovasc Pharmacol. 2011 Jan;57(1):86-93. doi: 10.1097/FJC.0b013e3181ffe8d0. PMID 20980920